CLINICAL TRIAL: NCT05496179
Title: The Effect of Prucalopride on Gastric Emptying in Intensive Care Unit Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Eman Mohamed El Mokadem, Lecturer of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Future University in Egypt
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Enteral Feeding Intolerance
MeSH Terms: interventions — prucalopride; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prucalopride (Active Comparator): Patients will receive prucalopride (2 mg) once daily for 7 days.
  Interventions: Drug: Prucalopride
- Metoclopramide (Active Comparator): Patients will receive metoclopramide (10 mg) three times daily for 7 days.
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Prucalopride — Prokinetic
  Other Names: Resolor
  Arms: Prucalopride
Drug: Metoclopramide — Prokinetic
  Other Names: Primperan
  Arms: Metoclopramide

SUMMARY:
to compare the effectiveness as well as the safety of prucalopride against metoclopramide as the first line treatment for feeding intolerance in critically ill patients.

DETAILED DESCRIPTION:
Provision of nutrition support to the critically ill is now established as an essential part of patient care where aiming toward 100% of the predicted target may have resulted in reduced mortality and increased ventilator-free days in those who are premorbidly malnourished. Despite these reported benefits, clinicians continue to deliver little more than half of the enteral nutrition (EN) they plan to provide, due to gastric motility disorders, patient intolerance and clinical interruptions. Also despite the availability of numerous clinical practice guidelines (CPGs) focused on feeding critically ill patients, observational studies have consistently demonstrated persistent and significant gaps between guideline recommendations and actual nutrition practice. Consequently, underfeeding is prevalent in the intensive care unit (ICU), with patients on average receiving only 60 % of the calories that are prescribed. Moreover, Among the barriers to adequate nutritional supply in the ICU which contributes to nutritional status deterioration, gastrointestinal disorders causing enteral feed intolerance are the most important and the most often mentioned in the literature. when gastric emptying was measured in critically ill patients, 46 % of them had evidence of delayed gastric emptying. Untreated slow gastric emptying has a plethora of clinical consequences such as vomiting, aspiration of gastric contents, pneumonia, and contributes significantly to the frequent interruptions and cessation of EN in the ICU, which results in inadequate nutritional delivery. Studies have shown an association between feeding intolerance, prolonged intensive care unit (ICU) stay, and increased risk of death.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging between 18 and 60 years (of both sexes) who are admitted to the ICU and are expected to stay in the ICU for not less than 7 days and are prescribed enteral feeding through naso- or oro-gastric tube whose modified nutritional risk in the critically ill (mNUTRIC) score is of more than or equal

Exclusion Criteria:

* Patients who met the following criteria were excluded:

  * Age less than 18 years or more than 60 years.
  * Previous upper gastrointestinal tract surgery, obstruction, hemorrhage or history of GI disease.
  * Clinically significant hepatic dysfunction. (>3 times above the upper end of normal range of bilirubin, γ-glutamyl transferase, aspartate transaminase, or lactate dehydrogenase)
  * Regular use of H2 blockers, prokinetic, proton pump inhibitor or anticholinergic agents for previous 4 weeks.
  * Patients with arrhythmia or atrioventricular blocks.
  * Any condition or comorbid disease that might interfere with gastric emptying such as diabetes.
  * Patients with head injuries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume | 7 days
  Gastric residual volume as a surrogate to gastric emptying by means of gastric residual volume

SECONDARY OUTCOMES:
Determining the adequacy of enteral nutrition: | 7 days
  Enteral nutrition volume ratio
Incidence of infectious complications. | one month
  C reactive protein
Length of ICU stay | 3 months
  duration of stay in intensive care unit
Adverse drug events | 7 days
  occurence of adverse drug events

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elmokadem, PhD, Principal Investigator — Future University in Egypt
Locations (1):
- Kasr Al Ainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elmokadem EM, Abou El Fadl DK, Eissa N, Alnassar NA, Bassiouny AM, Hanna Samy AE, El Said NO. Comparison of enteral prucalopride versus intravenous metoclopramide for feeding intolerance in patients with critical illness: a randomized double-blinded study. Front Pharmacol. 2024 Nov 8;15:1413246. doi: 10.3389/fphar.2024.1413246. eCollection 2024. PMID 39584139